CLINICAL TRIAL: NCT00080925
Title: T-Cell Depleted, Reduced-Intensity Allogeneic Stem Cell Transplantation From Haploidentical Related Donors For Hematologic Malignancies
Brief Title: T-Cell-Depleted Allogeneic Stem Cell Transplantation After Immunoablative Induction Chemotherapy and Reduced-Intensity Transplantation Conditioning in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 040116; 04-C-0116; CDR0000357432
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: prolymphocytic leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary acute myeloid leukemia; recurrent adult Hodgkin lymphoma; refractory anemia with excess blasts; refractory multiple myeloma; primary myelofibrosis; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; chronic myelomonocytic leukemia; polycythemia vera; essential thrombocythemia; stage II multiple myeloma; stage III multiple myeloma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Prolymphocytic; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Anemia, Refractory, with Excess of Blasts; Primary Myelofibrosis; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Leukemia, Myelomonocytic, Chronic; Polycythemia Vera; Thrombocythemia, Essential; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Filgrastim; Rituximab; Cyclophosphamide; Cyclosporine; Cytarabine; Doxorubicin; Etoposide; fludarabine phosphate; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: graft-versus-tumor induction therapy
Biological: rituximab
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: fludarabine phosphate
Drug: prednisone
Drug: vincristine sulfate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Donor peripheral stem cell transplantation may be able to replace bone marrow and immune cells that were destroyed by chemotherapy. Sometimes the transplanted cells from a donor are rejected by the body's normal cells. Eliminating the T cells from the donor cells before transplanting them and giving cyclosporine may prevent this from happening.

PURPOSE: This phase I trial is studying the side effects of T-cell-depleted allogeneic stem cell transplantation after immunoablative induction chemotherapy and reduced-intensity transplantation conditioning (chemotherapy) in treating patients with hematologic malignancies.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine engraftment in patients with hematologic malignancies treated with T-cell-depleted allogeneic stem cell transplantation after immunoablative induction chemotherapy and reduced-intensity transplantation conditioning.

Secondary

* Determine the incidence of acute graft-versus-host disease (GVHD), and nonrelapse mortality (within 100 days after transplantation) in these patients.
* Correlate levels of host immunosuppression before transplantation conditioning, as evaluated by peripheral blood CD4 counts, with graft rejection/failure within 100 days after transplantation and the level of donor hematopoietic chimerism 28 days after transplantation in these patients.
* Correlate donor-versus-recipient natural killer cell alloreactivity with graft rejection/failure, acute GVHD, and relapse of malignant disease in patients treated with this regimen.
* Determine the development of allospecific cytotoxic T-lymphocytes after transplantation in patients with myeloid or lymphoid leukemia.
* Correlate serum interleukin-7 and interleukin-15 levels with in vivo changes in host lymphocyte subpopulations in these patients during sequential immunoablative chemotherapy, before allogeneic stem cell transplantation, and during immune reconstitution after transplantation.

OUTLINE: This is a pilot study.

* Induction chemotherapy: Patients receive 1 of 2 induction chemotherapy regimens according to diagnosis. Patients with partial response or better after prior therapy (i.e., already adequately immune depleted) proceed directly to the transplantation preparative regimen.

  * Regimen A (Hodgkin's lymphoma, non-Hodgkin's lymphoma [except lymphoblastic lymphoma], chronic lymphocytic leukemia, prolymphocytic leukemia, or multiple myeloma): Patients receive rituximab IV (if they have CD20+ B-cell malignancies) on day 1; fludarabine IV over 30 minutes on days 1-4; etoposide, doxorubicin, and vincristine IV continuously on days 1-4; cyclophosphamide IV over 30 minutes on day 5; oral prednisone on days 1-5; and filgrastim (G-CSF) subcutaneously (SC) beginning on day 6 and continuing until blood counts recover.
  * Regimen B (lymphoblastic lymphoma, acute myeloid leukemia, acute lymphoblastic leukemia, refractory anemia with excess blasts, myeloproliferative disorders, chronic myelomonocytic leukemia, or chronic myelogenous leukemia): Patients receive G-CSF SC beginning 24 hours before initiating induction chemotherapy and continuing until blood counts recover. Patients also receive fludarabine IV over 30 minutes and cytarabine IV over 4 hours on days 1-5.

For both regimens, treatment repeats every 21 days for 1-2 courses. Patients who achieve remission or who have responsive or stable disease after induction chemotherapy then proceed to transplantation preparative regimen chemotherapy.

* Transplantation preparative regimen chemotherapy: Patients receive fludarabine IV over 30 minutes and cyclophosphamide IV over 2 hours on days -6 to -3.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours twice daily beginning on day -1 and continuing IV or orally until day 100. Patients with no acute GVHD at day 100 taper cyclosporine over 12 weeks.
* Allogeneic stem cell transplantation (SCT): Patients undergo T-cell-depleted allogeneic peripheral blood SCT on day 0. Patients receive G-CSF SC beginning on day 0 and continuing until blood counts recover.
* Donor lymphocyte infusion (DLI): Patients with persistent or progressive malignant disease after transplantation or mixed chimerism that does not improve after tapering or discontinuing immunosuppression therapy may receive DLI. DLI may be administered alone or in combination with chemotherapy. DLI repeats every 4 weeks until adequate donor chimerism is achieved or until GVHD develops.

Patients are followed at 28 and 100 days and then at 6, 9, 12, 18, and 24 months.

PROJECTED ACCRUAL: A total of 6-20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * In first complete remission (CR1), meeting 1 of the following criteria:

      * Adverse cytogenetics with minimal residual disease detectable by flow cytometry, cytogenetic analysis, fluorescence in situ hybridization (FISH), or polymerase chain reaction (PCR), defined as 1 of the following:

        * Complex karyotype [≥ 3 abnormalities]
        * inv(3) or t(3;3)
        * t(6;9)
        * t(6;11)
        * Monosomy 7
        * Trisomy 8, alone or with an abnormality other than t(8;21), t(9;11), inv(16), or t(16;16)
        * t(11;19) (q23;p13.1)
      * Failed to achieve CR after primary induction chemotherapy
      * Secondary AML
    * In second or subsequent remission (CR2 or greater)
  * Acute lymphoblastic leukemia, meeting 1 of the following criteria:

    * In CR1, meeting 1 of the following criteria:

      * Adverse cytogenetics with minimal residual disease detectable by flow cytometry, cytogenetic analysis, FISH, or PCR, defined as the following:

        * Translocations involving 11q23, t(9;22), or bcr-abl rearrangement
      * Failed to achieve CR after primary induction chemotherapy
    * In CR2, if CR1 was < 12 months
    * In CR3 or greater
  * Myelodysplastic syndromes (MDS)

    * INT-2 or high-risk by International Prognostic Scoring System
    * No MDS with Fanconi anemia
  * Chronic myelogenous leukemia (CML), meeting 1 of the following criteria:

    * Accelerated phase with treatment failure after imatinib mesylate
    * Blast phase
  * Myeloproliferative disorders, meeting 1 of the following criteria:

    * Agnogenic myeloid metaplasia with adverse-risk features, meeting at least 2 of the following criteria:

      * Hemoglobin < 10 g/dL or > 10g/dL if transfusion-dependent
      * WBC < 4,000/mm^3 OR > 30,000/mm^3 OR requires cytoreductive therapy to maintain WBC < 30,000/mm^3
      * Abnormal cytogenetics, including +8, 12p-
    * Polycythemia vera or essential thrombocythemia in transformation to secondary AML
  * Myelodysplastic/myeloproliferative disease

    * Chronic myelomonocytic leukemia
  * Hodgkin's lymphoma or non-Hodgkin's lymphoma

    * Refractory lymphoma with progressive disease during combination chemotherapy
    * Relapse after OR ineligible for autologous stem cell transplantation (SCT)
  * Chronic lymphocytic leukemia

    * Treatment failure* after fludarabine, chlorambucil, and at least 1 other salvage regimen
  * Prolymphocytic leukemia (PLL), meeting 1 of the following criteria:

    * T-PLL

      * Treatment failure* after alemtuzumab and at least 1 other regimen
    * B-PLL

      * Treatment failure* after fludarabine and at least 1 other salvage regimen
  * Multiple myeloma, meeting 1 of the following criteria:

    * Relapse after autologous SCT
    * Plasma cell leukemia
    * Adverse cytogenetics, defined as 1 of the following:

      * del(13q) = 11q translocation NOTE: *Treatment failure is defined as relapse within 6 months OR failure to achieve remission
* Less than 10% blasts in bone marrow and no circulating blasts in peripheral blood for the following diagnoses:

  * Primary or secondary leukemia
  * Refractory anemia with excess blasts
  * CML
  * Other eligible diagnosis in transformation to acute leukemia
* Expected survival of approximately 1 year or less with conventional therapy
* No active CNS involvement by malignancy*

  * Prior CNS involvement with no current evidence of CNS malignancy allowed NOTE: *Active CNS malignancy is defined by lymphoma: tumor mass on CT scan or leptomeningeal disease OR leukemia: blasts present on cerebrospinal fluid cytospin
* Availability of a donor who is a sibling, parent, or offspring who shares 1 full haplotype (HLA-A, -B, or -DR)

  * Recipient and donor must have at least a 2-antigen disparity in either the host-versus-graft or graft-versus-host direction
  * Parent or offspring donor who is mismatched for a single HLA antigen (i.e., 5/6 HLA) is allowed
  * No sibling donor who is 6/6 HLA-matched OR mismatched for a single HLA antigen (i.e., 5/6 HLA)
  * No unrelated donor identified in a prior or current National Marrow Donor Program registry search

PATIENT CHARACTERISTICS:

Age

* 18 to 55

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count ≥ 20,0000/mm^3* (without transfusion) NOTE: *Lower values may be accepted at the discretion of the principal investigator or study chairperson if due to bone marrow involvement by malignancy

Hepatic

* ALT and AST ≤ 2.5 times upper limit of normal (ULN)*
* Bilirubin ≤ 2.5 times ULN*
* Unconjugated hyperbilirubinemia consistent with Gilbert's syndrome allowed
* No chronic active hepatitis B infection

  * Hepatitis B core antibody positive allowed provided patient is surface antigen negative and has no evidence of active infection
* No hepatitis C viral infection

  * Seronegative for anti-hepatitis C antibody and detectable hepatitis C viral RNA by reverse transcriptase-polymerase chain reaction assay NOTE: *Higher levels may be accepted at the discretion of the principle investigator or study chairperson if such elevations are due to liver involvement by malignancy

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* LVEF ≥ 45%

Pulmonary

* DLCO ≥ 50% of expected value (corrected for blood hemoglobin level and alveolar volume)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study participation
* HIV negative
* No active infection not responding to antimicrobial therapy
* No psychiatric disorder that would preclude study compliance or informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 2 weeks since prior monoclonal antibody therapy

Chemotherapy

* See Disease Characteristics
* At least 2 weeks since prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from all prior therapy
* No administration of tyrosine kinase (TK) inhibitors, including imatinib mesylate and dasatinib, during the conditioning regimen; TK inhibitor administration may resume 28 days after transplantation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-02; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Bishop, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States